CLINICAL TRIAL: NCT06730425
Title: Examining Stress Salivary Biomarkers in Pediatric Patients Undergoing Dental Procedures. A Prospective Longitudinal Study
Brief Title: Examining Stress Salivary Biomarkers in Pediatric Patients Undergoing Dental Procedures
Status: Completed | Type: Observational
Sponsor: Midwestern University (Other)
Responsible Party: Sponsor
Other Study IDs: CIRB#IL24015
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Dental Anxiety; Dental Fear; Stress; Pediatric Population
Keywords: dental anxiety; pediatric patients; salivary biomarkers; salivary diagnostics; dental fear; stress; salivary cortisol; salivary alpha-amylase; salivary IgA

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Salivary sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric patients seen at the pediatric or orthodontic department: New pediatric patients seen for the first time at either the pediatric or the orthodontic department at the dental clinic of Midwestern University to start either a dental procedure or an orthodontic treatment

SUMMARY:
Pediatric patients are susceptible to show signs of fear. One of the scenarios that have always been a source of fear is undergoing a dental procedure. Fear of undergoing dental procedure has been addressed as "dental fear", which can lead to avoidance of receiving dental care and may result to a decline in proper oral hygiene.

Fear stimulates multiple cerebral responses and can be often related to an increased stress level. Stress level fluctuations during dental procedures can be examined by blood and salivary biomarkers. Given accessibility and minimal invasiveness, the collection of saliva samples constitutes an easy and cost-effective diagnostic method to investigate a variety of oral and systemic conditions. Cortisol and alpha amylase are present within the saliva and their levels are supposedly influenced by stress. In contrast, salivary IgA is not known to be influenced by stress level and can be used in comparison as a non-stress salivary biomarker.

Fear of dental appointments is a well-known cause of stress and activation of the sympathetic nervous system in adolescents undergoing dental procedure. However, the examination of stress and stress-related factors in young individuals attending their first dental appointment compared to young individuals who present for an orthodontic application is largely understudies.

Therefore, the aims of the study are: 1) to measure stress salivary biomarkers in pediatric patients before undergoing dental and/or orthodontic procedures; 2) assess whether subjective stress to dental treatment (as measured by dental anxiety, stress, and dental fear) is associated with objective stress measurements (as measured by collection of stress salivary biomarkers).

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 7 and 17
* Ability to read and speak English language
* Patients seen for a first visit at the pediatric or orthodontic departments of the dental institute of the Multispecialty Clinic at Midwestern University with a scheduled future appointment to start treatment in the pediatric or orthodontic department

Exclusion Criteria:

* Older than 17 years of age or younger than 7 years of age
* Unable to read and speak English language
* Have any major health conditions or history of mental illness
* Being a returning patient in the pediatric or orthodontic department of the dental institute of the Multispecialty Clinic at Midwestern University
* Taking any systemic medications that would cause a change in salivary flow (e.g., oxybutynin, protein pump inhibitors)

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: New pediatric patients that needs treatment at either the pediatric or the orthodontic departments of the dental institute at Midwestern University
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Correlation between psychological distress and levels of salivary biomarkers | At one time-point, before starting the dental procedure
  Levels of dental fear (measured with 15-75 Children's Fear Survey Schedule-Dental Subscale, with values >38 identifying dental fear), dental anxiety (measured with 8-40 Modified Child Dental Anxiety Scale, with values >19 identifying anxiety) and self-perceived stress (measured with 1-40 Perceived Stress Scale, with values >14 identifying stress) will be correlated with levels of salivary cortisol, alpha-amylase and IgA

CONTACTS AND LOCATIONS:
Locations (1):
- Midwestern University, Downers Grove, Illinois, United States